CLINICAL TRIAL: NCT02431741
Title: Title: A Prospective, Open, Non-controlled Clinical Investigation to Evaluate the Performance and Safety of an Antimicrobial Foam Transferring Dressing in Patients With Malignant Wounds
Brief Title: A Prospective, Open, Non-controlled Clinical Investigation to Evaluate the Performance and Safety of an Antimicrobial Foam Transferring Dressing in Patients With Malignant Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MxT Ag 03
Record Dates: First submitted 2015-04-28; First posted 2015-05-01 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2015-04

CONDITIONS: Malignant Wounds
Keywords: Presence of at least one exuding malignant (fungating) wound in need for antimicrobial treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mepilex Transfer Ag (Experimental): Non controlled investigation
  Interventions: Device: Mepilex Transfer Ag

INTERVENTIONS:
Device: Mepilex Transfer Ag

SUMMARY:
This is a prospective, open, non-controlled clinical investigation to evaluate the performance and safety of using Mepilex Transfer Ag on a malignant wound. Approximately ten to fifteen (10-15) subjects from one to three centers in Europe, presenting with a malignant (fungating) wound will be enrolled into the study. Eligible subjects will have one malignant (fungating) wound selected as a "study site". Subjects will be followed for a one-week observation period with their existing product followed by a 4-week investigation period using Mepilex Transfer Ag.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one exuding malignant (fungating) wound in need for antimicrobial treatment
* Both genders with an age ≥ 18 years at randomization
* Subjects with a suspected survival time of > 3 months
* Signed informed consent

Exclusion Criteria:

* Any known or suspected systemic infection
* Use of metronidazole is not allowed during the investigation period
* Any known sensitivity to silver or other components/products used in this study.
* Major uncontrolled systemic disorders such as hepatic, renal, neurologic, or endocrinologic disorders.
* Participation in another investigational study while participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Czechia (2):
  - Charles University School of Medicine, Prague, Prague
  - The General University Hospital in Prague, Prague, Prague

RESULTS

PARTICIPANT FLOW:
Groups:
- Mepilex Transfer Ag: Non controlled investigation
  Mepilex Transfer Ag
Period: Overall Study
Arm/Group | Mepilex Transfer Ag
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mepilex Transfer Ag
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 3
Region of Enrollment [Number; unit: participants]
  Czech Republic | 14
Infections in the wound at baseline [Number; unit: participants] — inclusion criteria is exuding malignant wound in need for antimicrobial treatment
  participants | 14
Pain during dressing changes [Number; unit: participants] | 14
Exudate handling [Number; unit: participants] — chronic wound exudate handling
  participants | 14
Presence of malodour [Number; unit: participants] | 14
Presence of bleeding from tumor [Number; unit: participants] | 14

OUTCOME MEASURES:

1. Primary Outcome: Infection in the Wound (Signs of Clinical Infection)
Description: Weekly Visual inspection of the wounds by the investigators.
Time Frame: weekly, for 5 weeks
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Mepilex Transfer Ag
Number analyzed (Participants) | 14
participants | 14

ADVERSE EVENTS:
Arm/Group | Mepilex Transfer Ag
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No